CLINICAL TRIAL: NCT06707194
Title: Effect and Safety of Benzathine Penicillin Combined With Etanercept on Spondyloarthritis: a Multicenter Randomized Controlled Clinical Study
Brief Title: Effect and Safety of Benzathine Penicillin Combined With Etanercept on Spondyloarthritis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NFEC-2025-283; NFSC-2024-060 (Other Grant/Funding Number: Southern Medical University, Nan Fang Hospital)
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Spondyloarthritis (SpA); Ankylosing Spondylitis (AS)
Keywords: spondyloarthritis; benzathine penicillin; Etanercept
MeSH Terms: conditions — Spondylarthritis; Spondylitis, Ankylosing | interventions — Etanercept; Penicillin G Benzathine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BPG with ETN (Experimental): Blinded "BPG with ETN" from Week 0 to Week 12, open-label "BPG with ETN" from Week 12 to Week 24.
  Interventions: Biological: Etanercept; Drug: Benzathine Penicillin
- Placebo with ETN (Placebo Comparator): Blinded "Placebo with ETN" from Week 0 to Week 12, open-label "BPG with ETN" from Week 12 to Week 24.
  Interventions: Biological: Etanercept; Drug: Benzathine Penicillin; Other: Placebo

INTERVENTIONS:
Biological: Etanercept — Prefilled syringe, 25mg of hypodermic injection, twice a week
Drug: Benzathine Penicillin — Preparation of suspension with appropriate amount of sterilized water (4-5ml) for injection, 1.2 million units of intramuscular injection, once every two weeks
Other: Placebo — Preparation of suspension with appropriate amount of sterilized water (4-5ml) for injection, intramuscular injection, once every two weeks
  Arms: Placebo with ETN

SUMMARY:
The purpose of the study is to verify the clinical feasibility of Benzathine penicillin (BPG) /Etanercept (ETN) combination regimen in patients with spondyloarthritis (SpA) and at the same time compare Benzathine penicillin /Etanercept combination regimen and Etanercept maintenance therapy in reducing disease activity, improving patients' clinical symptoms and body function scores, enhancing quality of life, improving imaging performance and safety.

DETAILED DESCRIPTION:
This trial is a randomised, double-blinded, placebo-controlled, polycentric study. The study consisted of a screening period (up to 2 weeks before randomization), a treatment period (24 weeks), and 5 follow-up visits (Weeks 0, 6, 12,18 and 24).

After a 2-week preparation period, 340 patients with SpA will be randomly and equally assigned to either experimental group consisting of BPG (injection form, 1.2 million units of intramuscular injection, once every two weeks) with ETN (injection form, 25mg of hypodermic injection, twice a week) or the control group consisting of placebos (injection form, once every two weeks) with ETN (injection form, 25mg of hypodermic injection, twice a week),with treatment lasting for 12 weeks. After 12 weeks of treatment, the label will be opened, and all patients will choose to use BPG combined with ETN maintenance therapy for another 12 weeks of treatment. Follow-up will be conducted at baseline, 6 weeks,12 weeks,18 weeks and 24 weeks after the end of treatment. The primary outcome is the response rate of ASAS40 in patients after 12 weeks of medication. The secondary outcomes are the severity of symptoms, disease activity, quality of life, and imaging progression scale scores of patients at each follow-up point. We will synchronize the recording of adverse events to compare the safety of the two treatment regimens

ELIGIBILITY:
Inclusion Criteria:

The following patients would be included: (1) The subjects voluntarily participate and sign an informed consent form; (2) patients aged 18-59 years; (3) According to the following guidelines or diagnostic criteria, a standardized diagnosis of spinal arthritis patients is made, which meets one of the following diagnostic criteria: ① 2009 ASAS classification criteria for axial spinal arthritis; ② Classification criteria for ASAS peripheral spondyloarthritis in 2011. And subjects with spinal arthritis who are in a relatively active period (ASDAS-CRP>1.2 )of infection;

Exclusion Criteria:

he exclusion criteria are as follows: (1) Subjects with nasopharyngitis, active tuberculosis, inflammatory bowel disease and other infections, other rheumatic and immune diseases, malignant tumors, and concomitant bone and joint diseases; (2) Individuals who are allergic to the components of the experimental drug; (3)Severe abnormalities in liver and kidney function (liver enzymes ≥ 2 times normal; creatinine ≥ 2 times normal); (4)Pregnant, preparing for pregnancy or breastfeeding women; (5)Moderate to severe heart failure (New York Heart Association grades 3-4); (6)Some researchers believe that other situations are not suitable for the use of etanercept or other experimental drugs; (7)Active gastrointestinal ulcer/bleeding; (8) According to the researcher's judgment, it is not suitable to participate in this study; (9)Patients in the acute phase of streptococcal infection: present with clinical manifestations of acute pharyngitis, acute tonsillitis, scarlet fever, and streptococcal pyoderma, and ASO or ADNS>normal range, and/or CRP>normal range.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-06-14 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Patient ASAS40 remission rate after 12 weeks of patient medication | Week 12
  Assessment of SpondyloArthritis International Society criteria (ASAS) consist of 4 domains measured on visual analog scales (VAS): 1. Patient's global assessment; 2. Patient's assessment of back pain; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). ASAS40 response is defined as an improvement of ≥40% and ≥2 units on a scale of 10 in at least three of the four ASAS main domains and no worsening at all in the remaining domain. A higher score on the VAS signifies higher severity.

SECONDARY OUTCOMES:
Improvement rate of Spondyloarthritis Research Consortium of Canada Score （SPARCC） | Baseline and Week 12、24
  The patients' sacroiliac joint MRIs were scored with reference to the Spondyloarthritis Research Consortium of Canada Score criteria, and the patients' pre-treatment scores were compared to calculate the rate of improvement
ASAS20 remission rate | Week 6、12、18、24
  Assessment of SpondyloArthritis International Society criteria (ASAS) consist of 4 domains measured on visual analog scales (VAS): 1. Patient's global assessment; 2. Patient's assessment of back pain; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). ASAS20 response is defined as an improvement of ≥20% and ≥1 units on a scale of 10 in at least three of the four ASAS main domains and no worsening at all in the remaining domain. A higher score on the VAS signifies higher severity.
Improvement rate of Spondyloarthritis Research Consortium of Canada Sacroiliac Joint Structural Score（SPARCCSSS） | Baseline and Week 12、24
  The patients' sacroiliac joint MRIs were scored with reference to the Spondyloarthritis Research Consortium of Canada Sacroiliac Joint Structural Score criteria, and the patients' pre-treatment scores were compared to calculate the rate of improvement
Change From Baseline in Patient Global Assessment | Baseline and Week 6、12、18、24
  Follow-up questionnaires were administered to the patients, including 1. average activity score of the spondylitis condition in the past week (0-10: never active to very active); 2. activity score of spondylitis in nocturnal pain (0-10: never active to very active)
Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index （BASDAI）Score | Baseline and Week 6、12、18、24
  Follow-up questionnaires were administered to patients, including: 1. overall degree of fatigue/drowsiness felt in the past week; 2. overall degree of neck, back, and hip pain felt in the past week; 3. overall degree of painful swelling in other joints (excluding neck, back, and hip pain) felt in the past week; 4. overall degree of discomfort felt in the past week due to touch or pressure; 5. overall degree of morning stiffness felt in the past week Overall degree of morning stiffness felt while awake; 6. Duration of morning stiffness when awake. Ranges from no impact (0 points) to very significant (10 points)
Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) Score | Baseline and Week 6、12、18、24
  Participants assessed their ability to perform 10 selected activities (e.g., putting on socks or tights without help or aids, bending forward from the waist to pick up a pen from the floor without an aid) during the preceding week. Responses ranged from 0 (easy) to 100 (impossible). The BASFI score is the average of the 10 responses and has a possible minimum value of 0 and a possible maximum value of 100.
C-reactive protein-based Ankylosing Spondylitis Disease Activity Score（ASDASCRP） | Baseline and Week 6、12、18、24
  0.121×total back pain+0.110×patient global+0.073×peripheral pain/swelling+0.058×duration of morning stiffness+0.579×Ln(CRP+1)
Change From Baseline in the scale of quality of life for ankylosing spondylitis (SQOL-AS) | Baseline and Week 6、12、18、24
  The scale consists of four areas: physiological functioning, psychological state, social functioning, and self-perception, with eight items to rate physiological functioning, six to rate psychological state, five to rate social functioning, and six to rate self-perception
Terms and Conditions for Using the 36-Item Short Form Survey（SF-36）（Physical Functioning (PF)、Mental Health (MH) ） | Baseline and Week 6、12、18、24
  The scale consists of two dimensions: physical functioning and mental health, with 10 items assessing physical functioning and 5 items assessing mental health.
Bath Ankylosing Spondylitis Metrology Index (BASMI) Score | Baseline and Week 12、24
  measure the lateral spinal flexion、tragus-to-wall distance、lumbar flexion (modified Schober)、maximal intermalleolar distance、cervical rotation
Change From Baseline in Maastricht ankylosing spondylitis enthesitis （MASES） score | Baseline and Week 12、24
  costochondral 1 right/left、costochondral 7 right/left、spina iliaca anterior superior right/left、crista iliaca right/left、spina iliaca posterior right/left、processus spinosus L5、achilles tendon, proximal insertion right/left. All sites are scored as 0 or 1. The MASES is the sum of all site scores (from 0 to 13)
Change From Baseline in Bath Ankylosing Spondylitis-Global （BAS-G） Score | Baseline and Week 6、12、18、24
  patient evaluation : 1. assess the impact of ankylosing spondylitis on health status in the past 1 week; 2. assess the impact of ankylosing spondylitis on health status in the past 6 months. (Scores range from 0 (none) to 10 (very severe).)
Change From Baseline in Work Productivity and Activity Impairment Specific Health Problem (WPAI-SHP) Questionnaire | Baseline and Week 6、12、18、24
  patient evaluation : 1. To what extent has the disease affected productivity while at work during the past seven days; 2. To what extent has the disease affected the ability to perform daily activities (other than work)? (Everyday activities are housework, shopping, child care, exercise, study, etc.) (Scores range from 0 (mild) to 10 (very severe))
Change From Baseline in Swollen Joint Count, Tender Joint Count | Baseline and Week 12、24
  Number of joints assessed by the patient for swelling and tenderness. All sites are scored as 0 or 1.
Change From Baseline in Indicators of streptococcal infection | Baseline and Week 6、12、18、24
  Patients had blood drawn for ASO, ADNase B, CRP, ESR indicators

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Nan Fang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia
  - Ganzhou People's Hospital, Ganzhou, Jiangxi

IPD SHARING:
Plan to Share IPD: Undecided